CLINICAL TRIAL: NCT03974022
Title: A Phase I/II, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of DZD9008 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) With EGFR or HER2 Mutation
Brief Title: Assessing an Oral EGFR Inhibitor, Sunvozertinib in Patients Who Have Advanced Non-small Cell Lung Cancer With EGFR or HER2 Mutation (WU-KONG1)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2019E0001
Record Dates: First submitted 2019-05-21; First posted 2019-06-04 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; EGFR; HER2; mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A Dose escalation (Experimental)
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 1 (Experimental)
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 2 (Experimental)
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 3 (Experimental): Patients with EGFR Exon20ins, previously treated with at least one line of systemic therapy
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 4 (Experimental): Patients with EGFR Exon20ins, previously treated with at least one line of systemic therapy
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 5 (Experimental): Patients with EGFR Exon20ins, treatment naïve
  Interventions: Drug: Sunvozertinib
- Part A Dose expansion cohort 6 (Experimental)
  Interventions: Drug: Sunvozertinib
- Part B Dose extension cohort 1 (Experimental): Patients with EGFR Exon20ins
  Interventions: Drug: Sunvozertinib
- Part B Dose extension cohort 2 (Experimental): Patients with EGFR Exon20ins
  Interventions: Drug: Sunvozertinib

INTERVENTIONS:
Drug: Sunvozertinib — Daily dose of Sunvozertinib
  Other Names: DZD9008

SUMMARY:
This study will treat patients with advanced NSCLC with EGFR or HER2 mutation who have progressed following prior therapy. This is the first time this drug is tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body and preliminarily assess its anti-cancer activity as monotherapy.

DETAILED DESCRIPTION:
A Phase I/II, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of Sunvozertinib in Patients with Advanced Non-Small Cell Lung Cancer (NSCLC) with EGFR or HER2 mutation. This study includes dose escalation, dose expansion, food effect (Part A) and dose extension (Part B).

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years old, be able to provide a signed and dated, written informed consent.
2. With documented histological or cytological confirmed locally advanced or metastatic NSCLC with EGFR or HER2 mutations.
3. (ECOG) performance status 0-1.
4. Predicted life expectancy ≥ 12 weeks
5. Patient must have measurable disease according to RECIST 1.1.
6. Patients with brain metastasis (BM) can be enrolled under the condition that BM is previously treated and stable, neurologically asymptomatic and does not require corticosteroid treatment.
7. Adequate organ system function.
8. Part A Dose expansion: Dose expansion cohort 5: NSCLC patients with EGFR Exon20ins, who have not received prior systemic therapy (treatment naïve).

   Part B Dose extension:
9. Patients must have histologically or cytologically confirmed locally advanced or metastatic NSCLC with documented EGFR Exon20ins mutation in tumor tissue from a local CLIA-certified laboratory (or equivalent) or Sponsor designated central laboratory prior to the study entry.
10. Patients should have received at least 1 line, but no more than 3 lines of systemic therapy for metastatic/locally advanced disease.

Exclusion Criteria:

1. For part B: Patients who have received prior treatment with Poziotinib or TAK788 or other EGFR/HER2 exon20 insertion inhibitors should be excluded. Prior treatment with currently approved EGFR TKIs for sensitizing or T790M resistance mutations, such as gefitinib, erlotinib, osimertinib, afatinib and dacomitinib, are allowed unless the patient had an objective response and subsequent progression assessed by the investigator.
2. Treatment with EGFR or HER2 antibodies, major surgery (excluding placement of vascular access), or onco-immunotherapy (e.g. immune checkpoint inhibitors PD-1, PD-L1, CTLA-4) within 4 weeks before the first administration of Sunvozertinib.
3. Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days before the first administration.
4. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose or with a wide field of radiation which must be completed within 4 weeks before the first administration.
5. Receiving (or unable to stop using) medications or herbal supplements known to be potent inhibitors or inducers of CYP3A within 1-2 weeks before the first administration.
6. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting Sunvozertinib with the exception of alopecia and grade 2 prior platinum-therapy related neuropathy.
7. Spinal cord compression or leptomeningeal metastasis.
8. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C, human immunodeficiency virus (HIV) and COVID-19 (per local practice).
9. Any of the following cardiac criteria: (1) Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs); (2) Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, and second-degree heart block, PR interval > 250 msec. (3) Any factors that increase the risk of QTF prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval; (4) Prior history of atrial fibrillation within 6 months of first administration of Sunvozertinib, except prior drug treatment related and recovered.
10. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
11. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Sunvozertinib.
12. History of hypersensitivity to active or inactive excipients of Sunvozertinib or drugs with a similar chemical structure or class to Sunvozertinib.
13. Women who are pregnant or breast feeding.
14. Involvement in the planning and conduct of the study.
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Antero Jänne, M.D & Ph. D, Principal Investigator — Dana-Farber Cancer Institute
Locations (124):
- United States (12):
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Orange, California
  - Innovative Clinical Research Institute, LLC, Whittier, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Northwell Health - Centers for Advanced Medicine, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (9):
  - Fundacion Respirar - Consultorios Medicos Dr. Doreski, Cabildo
  - CEMIC Centro de Educación Médica e Investigaciones Clínicas - Hospital Universitario sede Saavedra, Ciudad Autónoma Buenos Aires
  - Centro Medico Austral OMI, Ciudad Autónoma Buenos Aires
  - Diabaid, Ciudad Autónoma Buenos Aires
  - Fundacion CENIT Para La Investigacion en Neurociencias, Ciudad Autónoma Buenos Aires
  - Instituto Argentino de Diagnositco y Tratamiento S.A., Ciudad Autónoma Buenos Aires
  - Instituto Medico de la Fundacion de Estudios Clínicos, Ciudad Autónoma Buenos Aires
  - Centro de Investigación Pergamino SA, Pergamino
  - Clinica Viedma S.A, Viedma
- Australia (7):
  - Blacktown Hospital, Blacktown
  - Chris O'Brien Lifehouse, Camperdown
  - Austin Hospital, Heidelberg
  - St George Hospital, Kogarah
  - Peter MacCallum Cancer Centre - East Melbourne, North Melbourne
  - Linear Cancer trials, Perth
  - Southern Medical Day Care Centre, Wollongong
- Princess Margaret Cancer Centre, Toronto, Canada
- Chile (4):
  - Fundación Arturo López Pérez, Providencia
  - Orlandi Oncología - Centro Médico Health & Care, Santiago
  - SAGA, Santiago
  - James Lind Centro De Investigacion Del Cancer, Temuco
- China (33):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital，Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affilated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The first Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Henan Cancer Hospital, Henan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The Affiliated Huaian No.1 Peoples Hospital of Nanjing Medical University, Huai'an
  - Jinan Central Hospital, Jinan
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Medical University Cancer Hospital, Nanning
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- France (12):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron
  - Centre Georges François Leclerc, Dijon
  - CHU de Lille - Institut Coeur Poumons, Hellemmes-Lille
  - Hôpital de La Timone AP-Hm, Marseille
  - CHU de Montpellier Hôpital Arnaud de Villeneuve, Montpellier
  - APHP-Hôpital Bichat - Claude Bernard, Paris
  - CHU de Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - HIA Begin, Saint-Mandé
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - Institut Gustave ROUSSY, Villejuif
- Italy (9):
  - Centro di Riferimento Oncologico (CRO), Aviano
  - Azienda Ospedaliero - Universitaria "Policlinico - Vittorio Emanuele", Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST IRCCS, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - AUSL Romagna - Ospedale S.M delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituti Fisioterapici Ospitalieri, Roma
- Japan (6):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Tokushima University Hospital, Tokushima
  - Tokyo Shinagawa Hospital, Tokyo
- Malaysia (3):
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- South Korea (6):
  - Chungbuk National University Hospital, Cheonju
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (15):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - ICO (Institut Catala d'Oncologia) Badalona - Hospital Germans Trias i Pujol, Barcelona
  - Institut Català d'Oncología de Girona - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital de Jeréz, Jerez de la Frontera
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital La Fe, Valencia
- Taiwan (7):
  - Chi Mei Hospital, Liouying, Liuying
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Wan Fang Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang JC, Wang M, Doucet L, Fan Y, Lv D, Sun M, Huang D, Greillier L, Planchard D, Hong Q, Mazieres J, Felip E, Li X, Hu Y, Fang J, Bazhenova L, Ghiringhelli F, Cobo Dols MA, Rodriguez LP, Bearz A, Pellini B, Kim YJ, Bosch-Barrera J, Shim BY, Luo YH, Tiseo M, Yang TY, Carcereny E, Memmott RM, Zalcman G, de Castro Carpeno J, Di Noia V, Parra HS, Streich G, Lee DH, Shum E, Han JY, Jaime JC, Brungs D, John T, D'Arcangelo M, Joaquin AB, Liu G, Antonuzzo L, Hinojal GF, Le X, Zheng L, Janne PA; WU-KONG1B. Phase II Dose-Randomized Study of Sunvozertinib in Platinum-Pretreated Non-Small Cell Lung Cancer With Epidermal Growth Factor Receptor Exon 20 Insertion Mutations (WU-KONG1B). J Clin Oncol. 2025 Oct 10;43(29):3198-3208. doi: 10.1200/JCO-25-00788. Epub 2025 Sep 9. PMID 40923280
- [Derived] Luan T, Lin X, Xie X, Yang G, Wang S, Hao J, Zhou C. First case report of sunvozertinib for the treatment of HER2 exon 20 insertion in lung adenocarcinoma. Anticancer Drugs. 2024 Sep 1;35(8):757-760. doi: 10.1097/CAD.0000000000001628. Epub 2024 Jun 26. PMID 38924456

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 50 mg sunvozertinib, followed by a 7-day washout period. Then, they received sunvozertinib 50 mg once daily continuously.
- Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 100 mg sunvozertinib, followed by a 7-day washout period. Then, they received 100 mg sunvozertinib once daily continuously.
- Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 200 mg sunvozertinib, followed by a 7-day washout period. Then, they received 200 mg sunvozertinib once daily continuously.
- Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 300 mg sunvozertinib, followed by a 7-day washout period. Then, they received 300 mg sunvozertinib once daily continuously.
- Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 400 mg sunvozertinib, followed by a 7-day washout period. Then, they received 400 mg sunvozertinib once daily continuously.
- Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State: Patients with EGFR or HER2 exon20ins, previously treated with at least one line of systemic therapy.
  Patients received sunvozertinib 200 mg once daily dosing in the fasted state continuously.
- Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State: Patients with EGFR or HER2 exon20ins, previously treated with at least one line of systemic therapy.
  Patients received sunvozertinib 300 mg once daily dosing in the fasted state continuously.
- Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients received sunvozertinib 200 mg once daily dosing with a low-fat meal continuously.
- Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients received sunvozertinib 300 mg once daily dosing with a low-fat meal continuously.
- Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal: Patients with EGFR exon20ins, treatment naïve. Patients received sunvozertinib 300 mg once daily dosing with a low-fat meal continuously.
- Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg: Patients with EGFR exon20ins, were refractory to, relapsed from, or intolerant to previous amivantamab treatment.
  No patient was enrolled into this cohort.
- Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized at a 1:1 ratio to receive a single dose of sunvozertinib 300 mg under the High-Fat Meal condition, followed by a 7-day washout and crossed to receive a single dose of sunvozertinib 300 mg under the Fasted condition, followed by a 7-day washout. Then patients received sunvozertinib 300 mg once daily continuously.
- Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized at a 1:1 ratio to receive a single dose of sunvozertinib 300 mg under the Fasted condition, followed by a 7-day washout and crossed to receive a single dose of sunvozertinib 300 mg under the High-Fat Meal condition, followed by a 7-day washout. Then patients received sunvozertinib 300 mg once daily continuously.
- Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized to receive sunvozertinib 200 mg once daily continuously.
- Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized to receive sunvozertinib 300 mg once daily continuously.
Period: Overall Study
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Started | 3 | 6 | 3 | 7 | 6 | 10 | 14 | 14 | 7 | 31 | 0 | 5 | 7 | 91 | 111
Completed | 3 | 5 | 3 | 5 | 5 | 5 | 8 | 10 | 3 | 24 | 0 | 4 | 6 | 54 | 61
Not Completed | 0 | 1 | 0 | 2 | 1 | 5 | 6 | 4 | 4 | 7 | 0 | 1 | 1 | 37 | 50
Not completed — Death | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 33 | 40
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 2 | 3 | 0 | 1 | 0 | 3 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — site terminated by sponsor or non compliance | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patient was enrolled in Part A dose expansion cohort 6 due to conflict with enrollment of Part B.
Groups:
- Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 50 mg sunvozertinib, followed by a 7-day washout period. Then, they received 50 mg sunvozertinib once daily continuously.
- Total: Total of all reporting groups
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg | Total
Number analyzed (Participants) | 3 | 6 | 3 | 7 | 6 | 10 | 14 | 14 | 7 | 31 | 0 | 5 | 7 | 91 | 111 | 315
Age, Continuous [Median (Full Range); unit: years] | 48.0 [38 to 72] | 62.0 [48 to 83] | 57.0 [55 to 74] | 64.0 [57 to 82] | 63.5 [48 to 85] | 61 [41 to 83] | 62.5 [41 to 76] | 60.5 [34 to 73] | 64 [38 to 73] | 61 [37 to 96] |  | 44.0 [39 to 82] | 65.0 [55 to 78] | 62 [35 to 88] | 64 [37 to 89] | 62.0 [34 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 4 | 7 | 6 | 9 | 2 | 13 | 0 | 4 | 6 | 61 | 63 | 186
  Male | 0 | 3 | 1 | 4 | 2 | 3 | 8 | 5 | 5 | 18 | 0 | 1 | 1 | 30 | 48 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 5 | 2 | 5 | 3 | 10 | 9 | 13 | 7 | 23 | 0 | 1 | 0 | 59 | 65 | 204
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
  White | 1 | 1 | 1 | 2 | 3 | 0 | 5 | 1 | 0 | 5 | 0 | 4 | 6 | 30 | 44 | 103
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A Dose Escalation: Dose Limiting Toxicities (DLTs).
Description: To evaluate the safety and tolerability and defined the maximum tolerated dose (MTD) of sunvozertinib.
  DLT was evaluated in the DLT observation frame.
Time Frame: The DLT observation period is defined as the 28 days after the first multiple dose (up to 36 days from baseline).
Population: Patients in part A Dose Escalation Cohorts who met either or both criteria below were included in DLT analysis:
  * Patients who received the single dose and at least 80% of planned doses of DZD9008 in the first 28-day of repeated dosing and completed minimum required safety evaluations.
  * Patients who had at least one DLT reported during the DLT period. 1 patient in 100 mg dose level and 1 patient in 300 mg dose level received less than 80% of planned dose were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: Part B: Objective Response Rate (ORR) According to RECIST 1.1 by an Independent Review Committee (IRC).
Description: To evaluate anti-tumor activity of Sunvozertinib in advanced NSCLC patients with EGFR Exon20 insertion at defined dose(s) by assessment of Objective Response Rate (ORR).
Time Frame: through the study completion, an average of around 1 year for part B
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized ratio to receive sunvozertinib 300 mg once daily continuously.
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 85 | 107
percentage of participants | 45.9 [33.6 to 58.5] | 45.8 [34.8 to 57.0]
Statistical Analysis 1: Comparison: Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg; Test type: Superiority; p < 0.0001, binomial exact test against H0
Statistical Analysis 2: Comparison: Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg; Test type: Superiority; p < 0.0001, binomial exact test against H0

3. Secondary Outcome: Part B: DCR According to RECIST 1.1 Using Assessments Performed by an IRC; DCR Using Investigators Assessments According to RECIST 1.1
Description: To assess anti-tumor efficacy of Sunvozertinib using additional endpoints.
Time Frame: Through the study completion, an average of around 1 year for part B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized at a 1:1 ratio to receive sunvozertinib 200 mg once daily continuously.
- Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized at a 1:1 ratio to receive sunvozertinib 300 mg once daily continuously.
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 85 | 107
percentage of participants
  confirmed DCR by IRC | 89.4 [80.8 to 95.0] | 88.8 [81.2 to 94.1]
  confirmed DCR by investigator | 88.2 [79.4 to 94.2] | 88.8 [81.2 to 94.1]

4. Secondary Outcome: Part B: DoR, PFS According to RECIST 1.1 Using Assessments Performed by an IRC; DoR, PFS Using Investigators Assessments According to RECIST 1.1
Description: To assess anti-tumor efficacy of Sunvozertinib using additional endpoints.
Time Frame: Through the study completion, an average of around 1 year for part B
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 85 | 107
months
  Median duration of response (IRC) | NA [7.2 to NA] — NA means Not Estimable due to data not mature (lack of events observed being lower than 50%) | NA [6.7 to NA] — NA means Not Estimable due to data not mature (lack of events observed being lower than 50%)
  Median duration of response (investigator) | 8.3 [7.0 to NA] — NA means Not Estimable due to data not mature (lack of events observed being lower than 50%) | 8.8 [5.3 to 18.0]
  Median progression free survival (IRC) | 8.4 [6.8 to 11.2] | 6.9 [5.6 to 11.0]
  Median progression free survival (investigator) | 8.3 [5.5 to 10.9] | 6.8 [5.5 to 8.3]

5. Secondary Outcome: Part B: AEs/SAEs
Description: To determine the safety and tolerability of Sunvozertinib: Number of Participants With AEs, Number of Participants With SAEs. Using investigator reported AEs according to CTCAE and SAE criteria.
Time Frame: Through the study completion, an average of around 1 year for part B
Population: all patients had at least one dose of DZD9008
Measure: Number; unit: participants
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 91 | 111
participants
  Any TEAE | 91 | 111
  Any treatment- emergent SAE | 37 | 41

6. Secondary Outcome: Part A: Confirmed ORR and DCR by Investigator.
Description: To assess preliminary anti-tumor activity of sunvozertinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator.
  Confirmed ORR was defined as the percentage of patients achieving a CR (Complete Response) or PR (Partial Response) and was confirmed by subsequent tumor assessment at least 4 weeks within the study period.
  Confirmed DCR was defined as the proportion of patients with a best overall response of CR, PR, or SD. Patients who achieved a CR or PR must be confirmed by a subsequent tumor assessment at least 4 weeks within the study period.
  Patients who achieved a best overall response of SD must be confirmed by subsequent tumor assessment at least 35 days within the study period.
Time Frame: The study duration was from the initiation of sunvozertinib treatment until the study completion. The median study duration was 10 months, and the maximal study duration was 51.4 months for part A.
Population: Only participants in Part A were presented here, while Part B were presented separately. Participants in Part A with baseline and at least one post-treatment tumor assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 100 mg sunvozertinib, followed by a 7-day washout period. Then, they received sunvozertinib 100 mg once daily continuously.
- Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 200 mg sunvozertinib, followed by a 7-day washout period. Then, they received sunvozertinib 200 mg once daily continuously.
- Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 300 mg sunvozertinib, followed by a 7-day washout period. Then, they received sunvozertinib 300 mg once daily continuously.
- Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg: Patients with EGFR or HER2 mutations, previously treated with at least one line of systemic therapy.
  Patients received a single dose of 400 mg sunvozertinib, followed by a 7-day washout period. Then, they received sunvozertinib 400 mg once daily continuously.
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal
Number analyzed (Participants) | 3 | 6 | 3 | 7 | 5 | 10 | 13 | 14 | 5 | 29 | 0 | 5 | 7
percentage of participants
  Confirmed objective response rate | 0 [0.0 to 70.8] | 16.7 [0.4 to 64.1] | 0 [0.0 to 70.8] | 42.9 [9.9 to 81.6] | 0 [0.0 to 52.2] | 50 [18.7 to 81.3] | 30.8 [9.1 to 61.4] | 21.4 [4.7 to 50.8] | 40.0 [5.3 to 85.3] | 55.2 [35.7 to 73.6] |  | 20.0 [0.5 to 71.6] | 14.3 [0.4 to 57.9]
  Confirmed disease control rate | 100.0 [29.2 to 100.0] | 50.0 [11.8 to 88.2] | 66.7 [9.4 to 99.2] | 71.4 [29.0 to 96.3] | 60.0 [14.7 to 94.7] | 80 [44.4 to 97.5] | 84.6 [54.6 to 98.1] | 92.9 [66.1 to 99.8] | 80.0 [28.4 to 99.5] | 93.1 [77.2 to 99.2] |  | 60.0 [14.7 to 94.7] | 85.7 [42.1 to 99.6]

7. Secondary Outcome: Part A: DoR and PFS by Investigator.
Description: To assess preliminary anti-tumor activity of sunvozertinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator.
  DoR was presented for patients with confirmed objective response (CR or PR). DoR was the time from date of first documentation of CR or PR, which was subsequently confirmed, to date of first documentation of objective progression or death. Patients who had no documentation of objective progression or death was censored.
  PFS was the time from first dose date of sunvozertinib to date of first documentation of progression or death due to any cause, whichever occurred first. Patient who had no PFS event was censored.
Time Frame: The maximum median of DoR was 19.3 months, and the maximum median of PFS was 12.5 months for part A.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal
Number analyzed (Participants) | 3 | 6 | 3 | 7 | 5 | 10 | 13 | 14 | 5 | 29 | 0 | 5 | 7
month
  Median duration of response(month) | NA [NA to NA] — DoR cannot be calculated due to none achieved PR or CR. | 4.0 [NA to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | NA [NA to NA] — DoR cannot be calculated due to none achieved PR or CR. | 5.5 [2.8 to 5.5] | NA [NA to NA] — DoR cannot be calculated due to none achieved PR or CR. | NA [3.2 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 4.2 [3.2 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 6.3 [2.8 to 23.4] | 4.3 [3.0 to 5.6] | 9.8 [5.6 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). |  | 19.3 [NA to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 5.6 [NA to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%).
  Median progression free survival(month) | 3.1 [3.1 to 9.6] | 1.9 [0.9 to 22.5] | 12.5 [1.7 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 3.3 [1.2 to 7.4] | 4.6 [1.0 to 6.0] | 4.9 [1.2 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 5.5 [4.0 to 12.7] | 4.2 [2.4 to 9.0] | 4.2 [1.4 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%). | 10.8 [5.5 to 12.5] |  | 3.3 [1.4 to 21.3] | 5.3 [3.2 to NA] — NA means "not estimable" due to the data not being mature (i.e., the number of observed events is lower than 50%).

8. Secondary Outcome: Part A: Confirmed ORR and DCR by Independent Review Committee (IRC).
Description: To retrospectively assess anti-tumor activity of sunvozertinib in treatment-naive NSCLC patients with EGFR Exon20ins according to RECIST 1.1 by IRC.
  Confirmed ORR was defined as the percentage of patients achieving a CR or PR and was confirmed by subsequent tumor assessment at least 4 weeks within the study period.
  Confirmed DCR was defined as the proportion of patients with a best overall response of CR, PR, or SD. Patients who achieved a CR or PR must be confirmed by subsequent tumor assessment at least 4 weeks within the study period.
  Patients who achieved a best overall response of SD must be confirmed by subsequent tumor assessment at least 35 days within the study period.
Time Frame: as for outcome 6
Population: Only participants in Part A were presented here, while Part B were presented separately. According to the clinical study protocol, only participants in Part A Dose Expansion Cohort 5 (treatment-naive patients) were evaluated by IRC. Therefore, we only present the IRC results from Part A Dose Expansion Cohort 5.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal
Number analyzed (Participants) | 29
percentage of participants
  Confirmed objective response rate | 62.1 [42.3 to 79.3]
  Confirmed disease control rate | 89.7 [72.6 to 97.8]

9. Secondary Outcome: Part A Dose Escalation and Expansion: Maximum Plasma Concentration (Cmax) of DZD9008
Description: Maximum observed plasma concentration (ng/mL), obtained directly from the observed concentration versus time data. Calculated for the single dose.
Time Frame: Cycle 0 Day 1: 0 (predose) up to 168 hours (for Part A escalation); Cycle 1 Day 1: 0 (predose) up to 24 hours (for Part A expansion)
Population: All participants who have received at least one dose of study drug with at least one measurable plasma concentration of DZD9008 post dose without any important deviations or events that would exclude the participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg Daily: Patients with EGFR exon20ins, were refractory to, relapsed from, or intolerant to previous amivantamab treatment.
  No patient was enrolled into this cohort.
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg Daily
Number analyzed (Participants) | 3 | 6 | 2 | 7 | 4 | 10 | 10 | 13 | 7 | 29 | 0
ng/mL | 38.95 (37.3) | 89.19 (53.5) | NA (NA) — Not calculable, insufficient number of participants for calculation after excluding the data impacted by prohibited medication co-administration. | 428.8 (69.2) | 167.8 (90.7) | 176.3 (50.7) | 286.7 (62.6) | 253.0 (44.1) | 346.5 (33.5) | 354.3 (68.3) |

10. Secondary Outcome: Part A Dose Escalation and Expansion: Area Under the Plasma Concentration-time Curve From Zero to the Last Measurable Concentration (AUC0-t) of DZD9008
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear up/log down rule.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg
Number analyzed (Participants) | 3 | 6 | 2 | 7 | 4 | 10 | 10 | 13 | 7 | 29 | 0
h*ng/mL | 1434 (45.9) | 2693 (115.8) | NA (NA) — Not calculable, insufficient number of participants for calculation after excluding the data impacted by prohibited medication co-administration. | 12540 (69.7) | 6419 (60.0) | 2300 (46.0) | 3800 (56.9) | 3313 (39.3) | 4517 (28.2) | 4338 (60.3) |

11. Secondary Outcome: Part A Dose Escalation and Expansion: Cmax,ss, at Steady State of DZD9008
Description: Maximum observed plasma concentration(ng/mL), at steady state, obtained directly from the observed concentration versus time data. Calculated for the multiple dose.
Time Frame: Cycle 2 Day 1: 0 (predose) up to 24 hours (for Part A Dose expansion and expansion)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 3 | 9 | 10 | 9 | 4 | 19 | 0
ng/mL | 82.85 (17.2) | 229.4 (50.6) | NA (NA) — Not calculable, insufficient number of participants for calculation after excluding the data impacted by prohibited medication co-administration. | 590.2 (80.9) | 677.0 (21.9) | 358.0 (53.4) | 717.5 (40.9) | 613.3 (48.8) | 819.3 (57.3) | 716.5 (41.7) |

12. Secondary Outcome: Part A Dose Escalation and Expansion: AUCss, at Steady State of DZD9008
Description: Area under the plasma concentration-time curve in the dose interval at steady state, calculated by the linear up/log down rule.
Time Frame: Cycle 2 Day 1: 0 (predose) up to 24 hours (for Part A Dose escalation and expansion)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 3 | 9 | 10 | 9 | 4 | 19 | 0
h*ng/mL | 1506 (13.2) | 3823 (55.6) | NA (NA) — Not calculable, insufficient number of participants for calculation after excluding the data impacted by prohibited medication co-administration. | 10240 (78.1) | 12030 (25.2) | 5906 (52.3) | 11630 (40.3) | 9949 (45.8) | 14170 (47.9) | 12030 (40.2) |

13. Secondary Outcome: Part A Food Effect: Maximum Plasma Concentration (Cmax) of DZD9008
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data. Calculated for the single dose, in the fasted or fed state.
Time Frame: Day 1 and Day 9: 0 (predose) up to 168 hours.
Population: All participants from the food effect cohort for whom a PK profile is available on at least one of the fed and fasted dosing days.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A Food Effect Cohort: Sunvozertinib 300 mg: Patients with EGFR exon20ins, previously treated with at least one line of systemic therapy.
  Patients were randomized at a 1:1 ratio to receive a single dose of sunvozertinib 300 mg under the Fasted or High-Fat Meal condition, followed by a 7-day washout and crossed to receive a single dose of sunvozertinib 300 mg under the High-Fat Meal or Fasted condition, followed by a 7-day washout. Then patients received sunvozertinib 300 mg once daily continuously.
Arm/Group | Part A Food Effect Cohort: Sunvozertinib 300 mg
Number analyzed (Participants) | 12
ng/mL
  Part A Food effect: Maximum Plasma Concentration (Cmax) of DZD9008 under Fasted condition: number analyzed (Participants) | 11
  Part A Food effect: Maximum Plasma Concentration (Cmax) of DZD9008 under Fasted condition | 307.0 (59.6)
  Part A Food effect: Maximum Plasma Concentration (Cmax) of DZD9008 under High-Fat Meal condition | 331.6 (48.8)

14. Secondary Outcome: Part A Food Effect: Area Under the Plasma Concentration-time Curve From Zero to the Last Measurable Concentration (AUC0-t) of DZD9008
Description: Area under the plasma concentration-time-curve from time zero the last quantifiable time point, calculated by the linear up/log down rule, in the fasted or fed state.
Time Frame: Day 1 and Day 9: 0 (predose) up to 168 hours.
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A Food Effect Cohort: Sunvozertinib 300 mg
Number analyzed (Participants) | 12
h*ng/mL
  Part A Food effect: AUC0-t of DZD9008 under Fasted condition: number analyzed (Participants) | 11
  Part A Food effect: AUC0-t of DZD9008 under Fasted condition | 8266 (65.8)
  Part A Food effect: AUC0-t of DZD9008 under High-Fat Meal condition | 10050 (67.5)

15. Secondary Outcome: Part B: Maximum Plasma Concentration (Cmax) of DZD9008 and DZ0753
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data. Calculated for the single dose.
Time Frame: Cycle 1 Day 1: 0 (predose) up to 24 hours
Population: All dosed participants who have at least one measurable plasma concentration of DZD9008 post dose with no protocol deviations or adverse event thought to impact the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 22 | 21
ng/mL
  Part B: Maximum Plasma Concentration (Cmax) of DZD9008 | 173.4 (80.4) | 325.8 (73.7)
  Part B: Maximum Plasma Concentration (Cmax) of DZ0753 | 18.90 (113.4) | 40.40 (78.2)

16. Secondary Outcome: Part B: Area Under the Plasma Concentration-time Curve From Zero to the Last Measurable Concentration (AUC0-t) of DZD9008 and DZ0753.
Description: as for outcome 10
Time Frame: Cycle 1 Day 1: 0 (predose) up to 24 hours
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 22 | 21
h*ng/mL
  Part B: AUC0-t of DZD9008 | 2423 (71.9) | 4397 (55.7)
  Part B: AUC0-t of DZ0753 | 200.4 (125.2) | 448.5 (69.9)

17. Secondary Outcome: Part B: Cmax,ss, at Steady State of DZD9008 and DZ0753
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data. Calculated for the multiple dose.
Time Frame: Cycle 2 Day 1: 0 (predose) up to 24 hours
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 14 | 9
ng/mL
  Part B: Maximum Plasma Concentration (Cmax,ss) of DZD9008 | 342.8 (57.4) | 642.3 (48.1)
  Part B: Maximum Plasma Concentration (Cmax,ss) of DZ0753 | 42.58 (108.0) | 112.4 (83.7)

18. Secondary Outcome: Part B: AUCss, at Steady State of DZD9008 and DZ0753.
Description: Area under the plasma concentration-time curve from time zero in the dose interval at steady state, calculated by the linear up/log down rule.
Time Frame: Cycle 2 Day 1: 0 (predose) up to 24 hours
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
Number analyzed (Participants) | 14 | 9
h*ng/mL
  Part B: AUCss, at Steady State of DZD9008 | 6286 (56.1) | 10230 (47.5)
  Part B: AUCss, at Steady State of DZ0753 | 728.9 (112.2) | 1722 (84.9)

ADVERSE EVENTS:
Time Frame: Survival data continued to be collected for Part B participants following treatment discontinuation. SAEs and other AEs were monitored from the study treatment until the end of treatment, an average of approximately 11 months.
Description: No patient was enrolled in Part A dose expansion cohort 6 due to conflict with enrollment of Part B.
Arm/Group | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/6 | 0/3 | 2/7 | 0/6 | 1/10 | 0/14 | 2/14 | 1/7 | 4/31 | 0/0 | 0/5 | 0/7 | 33/91 | 40/111
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 1/3 | 4/7 | 2/6 | 4/10 | 5/14 | 9/14 | 2/7 | 14/31 | 0/0 | 0/5 | 1/7 | 37/91 | 41/111
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 7/7 | 6/6 | 10/10 | 14/14 | 14/14 | 7/7 | 31/31 | 0/0 | 5/5 | 7/7 | 91/91 | 111/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg (N=3) | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg (N=6) | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg (N=3) | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg (N=7) | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg (N=6) | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State (N=10) | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State (N=14) | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal (N=14) | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal (N=7) | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal (N=31) | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg (N=0) | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted (N=5) | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal (N=7) | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg (N=91) | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg (N=111)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anisocoria (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 6 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blue toe syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Escalation Cohort 1: Sunvozertinib 50 mg (N=3) | Part A Dose Escalation Cohort 2: Sunvozertinib 100 mg (N=6) | Part A Dose Escalation Cohort 3: Sunvozertinib 200 mg (N=3) | Part A Dose Escalation Cohort 4: Sunvozertinib 300 mg (N=7) | Part A Dose Escalation Cohort 5: Sunvozertinib 400 mg (N=6) | Part A Dose Expansion Cohort 1: Sunvozertinib 200 mg, Dosing in the Fasted State (N=10) | Part A Dose Expansion Cohort 2: Sunvozertinib 300 mg, Dosing in the Fasted State (N=14) | Part A Dose Expansion Cohort 3: Sunvozertinib 200 mg; Dosing With a Low-fat Meal (N=14) | Part A Dose Expansion Cohort 4: Sunvozertinib 300 mg; Dosing With a Low-fat Meal (N=7) | Part A Dose Expansion Cohort 5: Treatment naïve, Sunvozertinib 300 mg, Dosing With a Low-fat Meal (N=31) | Part A Dose Expansion Cohort 6: Previously Treated With Amivantamab; Sunvozertinib 300 mg (N=0) | Part A Food Effect Cohort 1: Sunvozertinib 300 mg; High-Fat Meal Condition First, Then Fasted (N=5) | Part A Food Effect Cohort 2: Sunvozertinib 300 mg; Fasted Condition First, Then High-Fat Meal (N=7) | Part B Dose Extension Cohort 1: EGFR exon20ins, Previously Treated; Sunvozertinib 200 mg (N=91) | Part B Dose Extension Cohort 2: EGFR exon20ins, Previously Treated; Sunvozertinib 300 mg (N=111)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 5 | 3 | 3 | 7 | 0 | 0 | 2 | 41 | 53
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 7
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 5 | 5
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 6 | 7
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 13 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 16 | 22
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 8
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 5 | 2 | 7 | 0 | 1 | 0 | 25 | 16
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 4 | 5 | 7 | 12 | 12 | 7 | 25 | 0 | 3 | 5 | 65 | 94
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 7 | 6
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 3
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 4 | 10
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 11 | 12
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3 | 2 | 7 | 6 | 3 | 5 | 0 | 4 | 4 | 28 | 48
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 4 | 4 | 10 | 0 | 0 | 0 | 18 | 22
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 5 | 1 | 6 | 3 | 1 | 7 | 0 | 0 | 1 | 32 | 49
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 13 | 30
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 3 | 6 | 1 | 5 | 0 | 2 | 3 | 24 | 22
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 5
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 10 | 4
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 4 | 14
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 5 | 0 | 1 | 2 | 7 | 10
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 7 | 8
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 9 | 15
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 7
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 2 | 1 | 2 | 2 | 4 | 6 | 7 | 2 | 17 | 0 | 2 | 0 | 26 | 43
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 9
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 9 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 1 | 0 | 20 | 18
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 4
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 4 | 0 | 2 | 1 | 12 | 17
Amylase increased (Investigations) | 0 | 0 | 1 | 4 | 1 | 1 | 1 | 2 | 1 | 6 | 0 | 0 | 2 | 16 | 18
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 5 | 0 | 2 | 1 | 18 | 19
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 7 | 6
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 14 | 0 | 0 | 1 | 35 | 59
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 4 | 5 | 0 | 2 | 2 | 26 | 35
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 11
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 6
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 6
Fluid balance negative (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid balance positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 7
Lipase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 6 | 0 | 1 | 3 | 21 | 17
Lung diffusion test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 10
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 12 | 16
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 5 | 12
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 3 | 0 | 1 | 0 | 23 | 28
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 12 | 11
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 3 | 1 | 1 | 4 | 5 | 4 | 11 | 0 | 2 | 1 | 44 | 45
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 1 | 8 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 14 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 2 | 0 | 2 | 1 | 19 | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 7 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 8 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 0 | 1 | 1 | 5 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 6
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 5 | 0 | 1 | 3 | 3 | 7
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 1 | 5 | 7
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 3 | 6 | 10
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 5 | 2 | 0 | 2 | 0 | 2 | 1 | 8 | 17
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 5
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meige's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 7
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 11 | 7
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 7
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 4 | 0 | 0 | 1 | 4 | 17
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 0 | 7 | 0 | 1 | 2 | 3 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 5 | 1 | 3 | 0 | 0 | 1 | 12 | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 4 | 0 | 0 | 0 | 7 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 7
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 0 | 3 | 2 | 2 | 7 | 0 | 0 | 2 | 7 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 2 | 4 | 4 | 1 | 8 | 0 | 1 | 1 | 19 | 29
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 8
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 4 | 1 | 6 | 0 | 0 | 0 | 24 | 26
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 3 | 1 | 4 | 6 | 1 | 16 | 0 | 1 | 0 | 34 | 52
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 5 | 3 | 4 | 3 | 7 | 0 | 2 | 0 | 6 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators, who are not employed by the sponsor, are free to publish study results. They must submit a copy of their publication to the sponsor for review at least 30 days in advance for manuscripts and 7 days for abstracts. The sponsor may request the removal of confidential information, identify patentable inventions, and provide comments. Publication may be delayed for up to 60 days to allow for a patent application. After this period, investigators can proceed with publication.

DOCUMENTS (2):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03974022/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT03974022/SAP_003.pdf